CLINICAL TRIAL: NCT01995370
Title: Cilostazol Stroke Prevention Study for Antiplatelet Combination
Acronym: CSPS・com
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Japan Cardiovascular Research Foundation (Other)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 021-TADD-1300-1; 000012180 (Other: UMIN)
Record Dates: First submitted 2013-11-15; First posted 2013-11-26 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Noncardioembolic Cerebral Infarction
Keywords: Noncardioembolic cerebral infarction; Dual antiplatelet therapy (DAPT); Cilostazol; Aspirin; Clopidogrel
MeSH Terms: interventions — Aspirin; Clopidogrel; Cilostazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Monotherapy group (Active Comparator): Aspirin (81mg or 100mg) or clopidogrel (50mg or 75mg) will be orally administered once daily.
  The treatment period will begin with the first visit of the first subject and end one year after the first visit of the last subject.
  Interventions: Drug: aspirin; Drug: clopidogrel
- DAPT group (Experimental): Cilostazol (100mg twice daily) will be orally administered in combination with aspirin (81 or 100mg once daily) or clopidogrel (50 or 75mg once daily).
  The treatment period will begin with the first visit of the first subject and end one year after the first visit of the last subject.
  Interventions: Drug: aspirin; Drug: clopidogrel; Drug: cilostazol

INTERVENTIONS:
Drug: aspirin — Aspirin (81mg or 100mg) will be orally administered once daily.The treatment period will begin with the first visit of the first subject and end one year after the first visit of the last subject.
  Other Names: Bayaspirin
Drug: clopidogrel — Clopidogrel (50mg or 75mg) will be orally administered once daily.The treatment period will begin with the first visit of the first subject and end one year after the first visit of the last subject.
  Other Names: Plavix
Drug: cilostazol — Cilostazol (100mg twice daily) will be orally administered. The treatment period will begin with the first visit of the first subject and end one year after the first visit of the last subject.
  Other Names: Pletaal OD Tablet
  Arms: DAPT group

SUMMARY:
To examine the efficacy and safety of dual antiplatelet therapy (DAPT) including cilostazol (Pletaal OD Tablet ®) in comparison with antiplatelet monotherapy (excluding cilostazol) for secondary prevention of ischemic stroke in high-risk patients for stroke

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of noncardioembolic IS that developed between 8 and 180 days before the start of the protocol treatment
* Patients with a responsible lesion identified by MRI
* Patients aged 20 to 85 years old when providing informed consent
* Patients taking clopidogrel or aspirin alone as antiplatelet therapy when providing informed consent
* Patients meeting at least one of the following criteria a-c:

  1. at least 50% stenosis of a major intracranial artery (to the level of A2, M2, or P2)
  2. at least 50% stenosis of an extracranial artery (the common carotid artery，internal carotid artery，vertebral artery，brachiocephalic artery，or subclavian artery)
  3. Two or more of the following risk factors

     * Aged 65 years or more
     * Diabetes mellitus
     * Hypertension
     * Peripheral arterial disease
     * Chronic kidney disease
     * History of IS (excluding the index IS for this study)
     * History of ischemic heart disease
     * Smoking (only current smokers)
* Patients considered to be able to visit the study site for ambulatory care throughout the observation period
* Patients who provided written informed consent

Exclusion Criteria:

* Patients with emboligenic heart disease
* Patients taking any anticoagulant agents
* Patients who cannot undergo MRI examination for reasons such as claustrophobia and implanted pacemaker
* Patients scheduled to undergo any surgery, such as percutaneous angioplasty, stent placement, and bypass grafting, during the study period
* Patients with a drug-eluting coronary stent implanted within one year
* Patients with a history of symptomatic non-traumatic intracranial hemorrhage, any other hemorrhagic disease (eg, active peptic ulcer), bleeding predisposition, or blood clotting disorders
* Patients with a history of hypersensitivity to cilostazol
* Patients with congestive heart failure or uncontrolled angina pectoris
* Patients with thrombocytopenia (platelet count ≦ 100,000/mm3)
* Patients with severe liver or renal dysfunction
* Women who are pregnant, breast-feeding, or of child-bearing potential
* Patients with a malignant tumor requiring treatment
* Patients who are taking aspirin, and meet any of the following criteria:

  * History of hypersensitivity to aspirin or salicylic acid analogues
  * Current peptic ulcer
  * Aspirin-induced asthma or its history
* Patients who are taking clopidogrel, and meet the following criterion:

  ・History of hypersensitivity to clopidogrel
* Patients who are participating in any other clinical studies
* Patients considered by the investigator/subinvestigator to be unsuitable for participating in this study

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1884 (Actual)
Dates: Start 2013-12-13 (Actual); Primary Completion 2018-12-07 (Actual); Study Completion 2018-12-07 (Actual)

PRIMARY OUTCOMES:
Recurrence of symptomatic ischemic stroke, with the symptoms lasting for at least 24 hours | every 6 months
  An "ischemic stroke" hereafter indicates a symptomatic ischemic stroke.

SECONDARY OUTCOMES:
Any stroke [ischemic stroke (IS), intracerebral hemorrhage (ICH), subarachnoid hemorrhage (SAH)] | every 6 months
SAH or ICH | every 6 months
IS or transient ischemic attack (TIA) | every 6 months
Death from any cause | every 6 months
Stroke (IS，ICH，SAH), myocardial infarction (MI), or vascular death | every 6 months
All vascular events: stroke, MI, and other vascular events | every 6 months
Adverse events and adverse drug reactions | every 6 months
Severe or life-threatening hemorrhage (GUSTO Criteria) | every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Takenori Yamaguchi, President emeritus, Principal Investigator — National Cerebral and Cardiovascular Center, Japan
Locations (1):
- Japan Cardiovascular Research Foundation, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koge J, Toyoda K, Koga M, Fukuda-Doi M, Uchiyama S, Kimura K, Hoshino H, Yamaguchi K, Okada Y, Sakai N, Miwa K, Minematsu K, Yamaguchi T; CSPS.com Trial Investigators. Effect of renal function on dual antiplatelet therapy using cilostazol for stroke prevention: a CSPS.com trial post hoc analysis. J Neurol Sci. 2025 Oct 15;477:123661. doi: 10.1016/j.jns.2025.123661. Epub 2025 Aug 18. PMID 40845415
- [Derived] Nishiyama Y, Kimura K, Otsuka T, Toyoda K, Uchiyama S, Hoshino H, Sakai N, Okada Y, Origasa H, Naritomi H, Houkin K, Yamaguchi K, Minematsu K, Matsumoto M, Tominaga T, Tomimoto H, Terayama Y, Yasuda S, Yamaguchi T; CSPS.com Trial Investigators. Dual Antiplatelet Therapy With Cilostazol for Secondary Prevention in Lacunar Stroke: Subanalysis of the CSPS.com Trial. Stroke. 2023 Mar;54(3):697-705. doi: 10.1161/STROKEAHA.122.039900. Epub 2023 Feb 3. PMID 36734235
- [Derived] Uchiyama S, Toyoda K, Okamura S, Omae K, Hoshino H, Kimura K, Kitagawa K, Minematsu K, Yamaguchi T. Dual antiplatelet therapy with cilostazol in stroke patients with extracranial arterial stenosis or without arterial stenosis: A subgroup analysis of the CSPS.com trial. Int J Stroke. 2023 Apr;18(4):426-432. doi: 10.1177/17474930221112343. Epub 2022 Jul 21. PMID 35762581
- [Derived] Toyoda K, Omae K, Hoshino H, Uchiyama S, Kimura K, Miwa K, Minematsu K, Yamaguchi K, Suda Y, Toru S, Kitagawa K, Ihara M, Koga M, Yamaguchi T; CSPS.com Trial Investigators. Association of Timing for Starting Dual Antiplatelet Treatment With Cilostazol and Recurrent Stroke: A CSPS.com Trial Post Hoc Analysis. Neurology. 2022 Mar 8;98(10):e983-e992. doi: 10.1212/WNL.0000000000200064. Epub 2022 Jan 24. PMID 35074890
- [Derived] Uchiyama S, Toyoda K, Omae K, Saita R, Kimura K, Hoshino H, Sakai N, Okada Y, Tanaka K, Origasa H, Naritomi H, Houkin K, Yamaguchi K, Isobe M, Minematsu K, Matsumoto M, Tominaga T, Tomimoto H, Terayama Y, Yasuda S, Yamaguchi T. Dual Antiplatelet Therapy Using Cilostazol in Patients With Stroke and Intracranial Arterial Stenosis. J Am Heart Assoc. 2021 Oct 19;10(20):e022575. doi: 10.1161/JAHA.121.022575. Epub 2021 Oct 8. PMID 34622679
- [Derived] Hoshino H, Toyoda K, Omae K, Ishida N, Uchiyama S, Kimura K, Sakai N, Okada Y, Tanaka K, Origasa H, Naritomi H, Houkin K, Yamaguchi K, Isobe M, Minematsu K, Matsumoto M, Tominaga T, Tomimoto H, Terayama Y, Yasuda S, Yamaguchi T; CSPS.com Trial Investigators. Dual Antiplatelet Therapy Using Cilostazol With Aspirin or Clopidogrel: Subanalysis of the CSPS.com Trial. Stroke. 2021 Nov;52(11):3430-3439. doi: 10.1161/STROKEAHA.121.034378. Epub 2021 Aug 18. PMID 34404237
- [Derived] Toyoda K, Uchiyama S, Yamaguchi T, Easton JD, Kimura K, Hoshino H, Sakai N, Okada Y, Tanaka K, Origasa H, Naritomi H, Houkin K, Yamaguchi K, Isobe M, Minematsu K; CSPS.com Trial Investigators. Dual antiplatelet therapy using cilostazol for secondary prevention in patients with high-risk ischaemic stroke in Japan: a multicentre, open-label, randomised controlled trial. Lancet Neurol. 2019 Jun;18(6):539-548. doi: 10.1016/S1474-4422(19)30148-6. PMID 31122494
- [Derived] Toyoda K, Uchiyama S, Hoshino H, Kimura K, Origasa H, Naritomi H, Minematsu K, Yamaguchi T; CSPS.com Study Investigators. Protocol for Cilostazol Stroke Prevention Study for Antiplatelet Combination (CSPS.com): a randomized, open-label, parallel-group trial. Int J Stroke. 2015 Feb;10(2):253-8. doi: 10.1111/ijs.12420. Epub 2014 Dec 8. PMID 25487817